CLINICAL TRIAL: NCT03937349
Title: Impact of Parathyroidectomy on Cardiovascular Calcification in Dialysis-dependent Patients: a Prospective Cohort Study
Brief Title: Impact of Parathyroidectomy on Cardiovascular Calcification in Dialysis-dependent Patients
Status: Completed | Type: Observational
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Ekaterina Parshina, Principal investigator, Saint Petersburg State University, Russia
Other Study IDs: Calcification
Record Dates: First submitted 2019-05-01; First posted 2019-05-03 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Secondary Hyperparathyroidism; Chronic Kidney Disease Mineral and Bone Disorder; Vascular Calcification; Dialysis
MeSH Terms: conditions — Hyperparathyroidism, Secondary; Chronic Kidney Disease-Mineral and Bone Disorder; Vascular Calcification

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sPTx group: Patients underwent subtotal parathyroidectomy due to severe secondary hyperparathyroidism
- TPTx+AT group: Patients underwent total parathyroidectomy with immediate autotransplantation of parathyroid tissue due to severe secondary hyperparathyroidism
- Control group: Patients with severe SHPT on conservative treatment (calcimimetics, active vitamin D analogues, phosphate-binders) who are likely to undergo surgery in a period of 12 months

SUMMARY:
This is a prospective cohort study aimed to evaluate change of cardiovascular calcification after parathyroidectomy in patients with end-stage renal disease on dialysis compared with control group on conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. ESRD patients receiving long-term hemodialysis or peritoneal dialysis treatment
3. Severe secondary hyperparathyroidism defined as iPTH level > 800 pg/ml, followed with hypercalcemia and/or hyperphosphatemia; with presence of one or more nodular or diffuse parathyroid hyperplasia confirmed with CT

Exclusion Criteria:

1. Primary hyperparathyroidosis as a cause of ESRD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving long-term dialysis treatment, met the criteria for parathyroidectomy due to severe SHPT
Sampling Method: Non-Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2024-01-18 (Actual); Study Completion 2024-01-18 (Actual)

PRIMARY OUTCOMES:
Change in coronary artery calcium score measured with CT | 18 months
Change in vascular calcification score measured with semi-quantitative (Kauppila) test | 18 months

SECONDARY OUTCOMES:
Change in heart valve calcium score | 18 months
Change in intact parathyroid hormone (iPTH) level | 18 months
Change in serum calcium level | 18 months
Change in serum phosphate level | 18weeks
Change in alkaline phosphatase | 18 months
Serious adverse events (cardiovascular events, death, fractures, emergency hospital admissions) during the follow-up period | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ekaterina Parshina, MD, Principal Investigator — Saint Petersburg State University, Russia
Locations (1):
- Saint-Petersburg State University, Clinic of advanced medical technologies n.a. N.I.Pirogov, Saint Petersburg, Russia